CLINICAL TRIAL: NCT06760039
Title: Safety and Efficacy of R-CMOP Versus R-CHOP in the Initial Treatment of Low-risk and Medium-risk Diffuse Large B-cell Lymphoma (DLBCL): a Randomized, Controlled, Open-label, Multicenter, Phase Ib/II Clinical Study
Brief Title: Safety and Efficacy of R-CMOP Versus R-CHOP in the Initial Treatment of DLBCL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-737-01
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; R-CHOP; Liposomal Mitoxantrone
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): R-CMOP group
  Interventions: Drug: R-CMOP Regimen
- Control group (Active Comparator): R-CHOP group
  Interventions: Drug: R-CHOP Regimen

INTERVENTIONS:
Drug: R-CMOP Regimen — Rituximab intravenous drip, Cyclophosphamide intravenous drip, Liposomal Mitoxantrone intravenous drip, Vincristine intravenous drip, Prednisone orally
  Arms: Experimental group
Drug: R-CHOP Regimen — Rituximab intravenous drip, Cyclophosphamide intravenous drip, Doxorubicinin intravenous drip, Vincristine intravenous drip, Prednisone orally
  Arms: Control group

SUMMARY:
This is a prospective, randomized, controlled, multicenter, phase II clinical trial to evaluate the efficacy and safety of R-CMOP versus R-CHOP in the initial treatment of low-risk and medium-risk diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged ≥18,≤80 years, both male and female.
2. Pathologically confirmed DLBCL
3. No prior treatment for DLBCL.
4. There must be at least one measurable or evaluable lesion that meets the evaluation criteria for Lugano 2014 lymphoma.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-
6. Expected survival ≥3 months.
7. International Prognostic Index (IPI) ≤ 2
8. Sufficient bone marrow, liver, and kidney function.

Key Exclusion Criteria:

1. Other types of LBCL:Primary Cutaneous Diffuse Large B-cell Lymphoma (Leg Type), Primary Mediastinal (Thymic) Large B-cell Lymphoma, Lymphomatoid Granulomatosis, ALK-positive Diffuse Large B-cell Lymphoma, Plasmablastic Lymphoma, Intravascular Large B-cell Lymphoma, T-cell/Histiocyte-rich Large B-cell Lymphoma, and others.
2. Transformed DLBCL.
3. Patients with central nervous system involvement, or those who require high-dose methotrexate for prevention.
4. The patients had previously received antitumor therapy.
5. Patients with the infection of human immunodeficiency virus (HIV) and/or acquired immunodeficiency syndrome.
6. Pregnant and lactating women and subjects of childbearing age who do not want to use contraception.
7. Mentally ill persons or persons unable to obtain informed consent.
8. The investigators think that the patient is not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
2-year event-free survival (EFS) rate assessed by the independent review committee | Defined as the proportion of patients without disease progresion, treatment discontinuation, or death for any reason within 24 months of enrollment, based on the independent review committee's assessment.
  To investigate the antitumor efficacy
RP2D(Phase Ib) | Cycle 1 in R-CMOP group (28 days)
  Phase II Recommended Dose
DLT(Phase Ib) | Cycle 1 in R-CMOP group (28 days)
  Dose-limiting toxicity

SECONDARY OUTCOMES:
2-year event-free survival (EFS) rate assessed by the investigators | Defined as the proportion of patients without disease progresion, treatment discontinuation, or death for any reason within 24 months of enrollment, based on the investigators' assessment.
  To investigate the anti-tumor efficacy
AE and SAE (Phase Ib) | Up to 24 weeks
  Number of participants with adverse events (AE) and severe adverse events (SAE) in phase Ib
2-year Progression-free survival(PFS) | Defined as the proportion of patients without disease progresion, treatment discontinuation, or death for any reason within 24 months of enrollment
  To investigate the antitumor efficacy
2-year Overall survival(OS) | Defined as the proportion of patients without disease progresion, treatment discontinuation, or death for any reason within 24 months of enrollment
  To investigate the antitumor efficacy
Objective response rate (ORR) | Up to 24 weeks
  To investigate the antitumor efficacy
Complete response rate (CRR) | Up to 24 weeks
  To investigate the antitumor efficacy

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - The Fifth Affiliated Hospital of Guangzhou Medical University., Guangzhou, Guangdong
  - The Affiliated Hospital of Guangdong Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Guangxi Zhuang Autonomous Region Cancer Hospital, Guilin, Guangxi
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - Beijing Tongren Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided